CLINICAL TRIAL: NCT00669487
Title: A 72-week Randomized Clinical Trial Comparing the Safety and Efficacy of Three Initial Antiretroviral Regimens -GPO-VIR S (d4T/3TC/NVP) for 24 Weeks Followed by GPO-VIR Z (AZT/3TC/NVP) vs GPO-VIR Z vs TDF/FTC/NVP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: Queen Savang Vadhana Memorial Hospital, Thailand (Other); Thai Red Cross AIDS Research Centre (Other); University of Hawaii (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Jintanat Ananworanich, SEARCH Research Foundation
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SEARCH003
Record Dates: First submitted 2008-04-24; First posted 2008-04-30 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections
Keywords: HIV/AIDS patients
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. GPO-VIR S 1 pill orally every 12 hours (Experimental)
  Interventions: Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP
- 2 GPO-VIR Z 1 pill orally every 12 hours (Experimental)
  Interventions: Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP
- 3 Truvada 1 pill oral q 24 hr and NVP 1 pill oral q 12 hr (Experimental)
  Interventions: Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP

INTERVENTIONS:
Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP — Truvada(FTC200mg+TDF300mg) every 24 hours + NVP 200 mg every 12 hours orally until week 72
  Arms: 3 Truvada 1 pill oral q 24 hr and NVP 1 pill oral q 12 hr
Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP — GPO-VIR S(D4T30mg+3TC150mg+NVP200mg)1 pill orally every 12 hours until week 24 and then switch to GPO-VIR Z
Drug: AZT/3TC/NVP, AZT/D4T/NVP, Truvada/NVP — GPO-VIR Z(AZT250mg+3TC150mg+NVP200mg) 1 pill orally every 12 hours until week 72

SUMMARY:
This protocol aims to determine the risk/benefits of this policy by comparing head-to-head a regimen of GPO-VIR Z or TDF/FTC/NVP for 18 months in ARV-naïve patients to a 6-month lead in with GPO-VIR S followed by 12 months of GPO-VIR Z. The primary outcomes to be assessed will be anemia, neuropathy, lipoatrophy and renal function.

DETAILED DESCRIPTION:
GPO-VIR Z is a new combination antiretroviral (ARV) medication that substitutes zidovudine (AZT) for stavudine (d4T) from the original formulation of GPO-VIR S. This new combination should decrease rates of lipoatrophy and neuropathy which are side-effects strongly linked to the use of d4T. However, there is some risk that initiating therapy with an AZT- containing regimen may cause unacceptable rates of anemia. Many Thai physicians have adopted a practice of using 6 months of the stavudine-containing GPO-VIR S as a lead in before introducing AZT-containing GPO-VIR Z in an effort to balance the risks and benefits of these two medications. There are no definitive data, however, that can attest to the benefit of such an approach.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection
2. Age ≥ 18 years old.
3. Subjects must be naïve to ARV. Individuals with past exposure to ARV associated with pregnancy will be allowed to enroll as long as the exposure is at least 3 months prior to entry.
4. CD4 < 350 cells/mm3
5. Subject understands the study and is able to sign informed consent

Exclusion Criteria:

1. Evidence of symptomatic persistent symptoms of tingling or numbness of lower extremities and bilateral lower extremity neuropathy on exam at entry. Abnormal exam includes 1) Diminished (compared with the knee) or absent ankle reflexes OR 2) Diminution of either vibration sensation in the legs (defined as perception of vibration for < 10 seconds at the great toe with a tuning fork initially struck hard enough to be audible) OR 3) Diminution of pin or temperature sensation in lower extremities OR 4) Contact allodynia in the feet.
2. Laboratory values 1) Absolute neutrophil count (ANC) < 750/mm3 2) Hemoglobin < 8.0 g/dL 3) ALT (SGPT) > 5 x ULN 4) Creatinine > 2 X ULN or < creatinine clearance < 30 cc per min by Cockroft-Gault formula
3. Active AIDS-defining opportunistic infection (OI) within 30 days prior to entry. Subjects must be off all acute treatments for OI for at least 14 days prior to entry. Subjects on maintenance or prophylactic therapy for AIDS-related OIs will be eligible.
4. Any immunomodulator, HIV vaccine or investigational therapy within 30 days of study entry
5. Pregnancy or breast-feeding; intent to become pregnant during the course of the study.
6. Presence of any active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean hemoglobin at 24 weeks and 72 weeks | 72 weeks
Proportion of participants with peripheral neuropathy at 24 weeks and 72 weeks | 72 weeks

SECONDARY OUTCOMES:
Changes from baseline in body weight, limb fat, and lean body mass by DEXA scan at 24 weeks and 72 weeks | 72 weeks
Change from baseline in serum creatinine at 24 weeks and 72 weeks | 72 weeks
Proportion of participants with plasma HIV-1 RNA less than 50 copies/mL at 24 weeks and 72 weeks | 72 weeks
Change from baseline in CD4 count at 24 weeks and 72 weeks | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat - Ananworanich, M.D., Principal Investigator — SEARCH Thailand; Jintanat - Ananworanich, M.D., Ph.D, Principal Investigator — SEARCH Thailand
Locations (1):
- SEARCH Thailand, Bangkok, Bangkok, Thailand